CLINICAL TRIAL: NCT02624336
Title: Evaluation of Synergistic Anti-plaque Activity of Salvadora Persica L. and Green Tea: A Clinical Comparative Study
Acronym: ESAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 101269-2
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
Keywords: periodontal disease; caries
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DTC1 mouth wash (Active Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: DTC1
- Oradex mouth wash (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Oradex
- Distilled water (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Distilled water

INTERVENTIONS:
Other: DTC1 — 15ml DTC1 twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: DTC1 mouth wash
Other: Oradex — 15ml Chlorhexidine gluconate 0.12% (w/v) twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Other Names: CHX
  Arms: Oradex mouth wash
Other: Distilled water — 15ml distilled water twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Distilled water

SUMMARY:
Accumulation of dental plaque may result in negative effects on the tooth and tooth supporting periodontal tissue. In addition, it contributes to the development of caries and periodontal diseases. Therefore, an effective dental plaque control is essential for maintaining good oral hygiene. Mechanical plaque control has its limitation thus chemical plaque control may be used as an adjunct in dental plaque control. Various types of medicinal plants can be utilized as stable, safe and biologically active plant-derived galenicals as alternative to synthetic mouth wash. Among these plants, Salvadora persica L. (Sp) root sticks and green tea (Gt) aqueous extracts were reported to have anti-microbial activity against many oral bacteria. The objective of this study was to investigate the efficacy of the combination of Gt aqueous extract and Sp aqueous extract as a synergistic anti-bacterial and anti-adherence efficacy against primary plaque colonizers.

DETAILED DESCRIPTION:
Dental plaque is the soft deposits that form the biofilm adhering to the tooth surface or other hard surfaces inside oral cavity, including removable and fixed restoration. The dental plaque is composed of over 500 bacterial species. The colonization of these bacteria follows a special pattern starting by adhesion of initial bacterial colonizers to the salivary pellicles covering tooth enamel and other hard surfaces in the oral cavity followed by secondary colonization of follower bacteria through inter-bacterial adhesion leading to dental plaque maturation.

Periodontal health can be considered to be in a state of balance when the bacterial mass presents in the host oral cavity and causes no damage to either the bacteria or the host periodontal tissues. Any disruption of this balance results in alterations in both the host periodontal and biofilm bacteria and leads ultimately to destruction of the periodontium. Accumulation of dental plaque may lead to several harmful effects on the tooth and tooth supporting periodontal tissue that contributes to the development of caries and periodontal diseases. Therefore, an effective dental plaque control is essential for maintaining good oral hygiene.

Mechanical plaque control, by using toothbrushes and interdental aids, is the mostly adopted method. Unfortunately, it is a time consuming process and needs high manual dexterity. Moreover, epidemiological studies revealed high prevalence of gingivitis among toothbrush users. Hence, chemical plaque control may be used to assist in dental plaque control.

The anti-plaque agent is that agent that interferes with one of the different phases of dental plaque development: interferes with the adhesion of oral bacteria to oral surfaces and prevent biofilm formation; interferes with co-aggregation mechanism which thereby prevents future growth of micro-colonies; or removes or disrupts existing dental plaque. To date, chlorhexidine (CHX) mouthwash is the standard solution used in chemical plaque control, but it was found to have several side effects including tooth and some restorations staining, unpleasant test, sloughing of oral mucosa and enhancement of supra-gingival calculus formation.

The widely available traditional natural medicinal plants can be utilized as stable, safe and biologically active plant-derived galenicals as alternative to synthetic drugs. Among these plants, Salvadora persica L. (Sp) root sticks and green tea (Gt), leafs of Camellia sinensis. Kuntze, aqueous extracts were reported to have anti-microbial activity against many oral bacteria. In our in vitro study, we found that the combination (Co.) of 0.25mg Gt aqueous extract and 7.82mg Sp aqueous extract in 1ml exhibited significant synergistic anti-bacterial and anti-adherence efficacy against primary plaque colonizers.

The dental plaque is classified into two categories, supra-gingival plaque and sub-gingival plaque, in relation to gingival margin. The supra-gingival dental plaque may be readily visualized on teeth after 24 to 48 hours with no oral hygiene measures and it appears white, grayish, or yellow in color and has a globular appearance.

Supra-gingival plaque accumulation on tooth surfaces can be quantified through different plaque index systems. In this study, the clinical parameter to record plaque quantity was modified Quigely Hein Plaque Index. In this index, a score of 0 to 5 was assigned for each facial and lingual (palatal) surface of all teeth except the third molars.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be medically healthy.
* Participants should have more than 20 teeth.

Exclusion Criteria:

* Participants who have active cavity caries and/or periodontal disease.
* Participants who have ongoing orthodontic treatment.
* Participants who have been on antibiotics within the past 4 months.
* Participants who require prophylactic antibiotic coverage.
* Participants who have been on systemic or topical non-steroidal anti-inflammatory drugs for the past 4 months.
* Participants who are pregnant or intended to and lactating mother.
* Participants who have heart valve replacement and have known intolerance or allergy to mouth rinses.
* Participants who have any systemic disease.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mean amount plaque between different DTC1 and placebo comparators i.e. Oradex and distilled water, as anti-plaque agent following 24 hrs plaque regrowth clinical trial by means of modified Quigely Hein Plaque Index [Turesky, 1970]. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nor_Adinar Baharuddin, DClinDent, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addy M, Moran J, Newcombe R, Warren P. The comparative tea staining potential of phenolic, chlorhexidine and anti-adhesive mouthrinses. J Clin Periodontol. 1995 Dec;22(12):923-8. doi: 10.1111/j.1600-051x.1995.tb01796.x. PMID 8613560
- [Background] Allison DG, Gilbert P. Modification by surface association of antimicrobial susceptibility of bacterial populations. J Ind Microbiol. 1995 Oct;15(4):311-7. doi: 10.1007/BF01569985. PMID 8605070
- [Background] Baehni PC, Takeuchi Y. Anti-plaque agents in the prevention of biofilm-associated oral diseases. Oral Dis. 2003;9 Suppl 1:23-9. doi: 10.1034/j.1601-0825.9.s1.5.x. PMID 12974527
- [Background] Chelli-Chentouf N, Tir Touil Meddah A, Mullie C, Aoues A, Meddah B. In vitro and in vivo antimicrobial activity of Algerian Hoggar Salvadora persica L. extracts against microbial strains from children's oral cavity. J Ethnopharmacol. 2012 Oct 31;144(1):57-66. doi: 10.1016/j.jep.2012.08.025. Epub 2012 Aug 29. PMID 22963838
- [Background] Dhar V, Jain A, Van Dyke TE, Kohli A. Prevalence of gingival diseases, malocclusion and fluorosis in school-going children of rural areas in Udaipur district. J Indian Soc Pedod Prev Dent. 2007 Apr-Jun;25(2):103-5. doi: 10.4103/0970-4388.33458. PMID 17660647
- [Background] Farnsworth NR, Akerele O, Bingel AS, Soejarto DD, Guo Z. Medicinal plants in therapy. Bull World Health Organ. 1985;63(6):965-81. PMID 3879679
- [Background] Hellden L, Camosci D, Hock J, Tinanoff N. Clinical study to compare the effect of stannous fluoride and chlorhexidine mouthrinses on plaque formation. J Clin Periodontol. 1981 Feb;8(1):12-6. doi: 10.1111/j.1600-051x.1981.tb02019.x. PMID 7019266
- [Background] Ismail AI, Szpunar SM. The prevalence of total tooth loss, dental caries, and periodontal disease among Mexican Americans, Cuban Americans, and Puerto Ricans: findings from HHANES 1982-1984. Am J Public Health. 1990 Dec;80 Suppl(Suppl):66-70. doi: 10.2105/ajph.80.suppl.66. PMID 9187585
- [Background] Manganiello AD, Socransky SS, Smith C, Propas D, Oram V, Dogon IL. Attempts to increase viable count recovery of human supragingival dental plaque. J Periodontal Res. 1977 Mar;12(2):107-19. doi: 10.1111/j.1600-0765.1977.tb00113.x. No abstract available. PMID 138728
- [Background] Rosan B, Lamont RJ. Dental plaque formation. Microbes Infect. 2000 Nov;2(13):1599-607. doi: 10.1016/s1286-4579(00)01316-2. PMID 11113379
- [Background] Sofrata A, Brito F, Al-Otaibi M, Gustafsson A. Short term clinical effect of active and inactive Salvadora persica miswak on dental plaque and gingivitis. J Ethnopharmacol. 2011 Oct 11;137(3):1130-4. doi: 10.1016/j.jep.2011.07.034. Epub 2011 Jul 20. PMID 21798329
- [Background] Sofrata A, Santangelo EM, Azeem M, Borg-Karlson AK, Gustafsson A, Putsep K. Benzyl isothiocyanate, a major component from the roots of Salvadora persica is highly active against Gram-negative bacteria. PLoS One. 2011;6(8):e23045. doi: 10.1371/journal.pone.0023045. Epub 2011 Aug 1. PMID 21829688
- [Background] Teles RP, Teles FR. Antimicrobial agents used in the control of periodontal biofilms: effective adjuncts to mechanical plaque control? Braz Oral Res. 2009;23 Suppl 1:39-48. doi: 10.1590/s1806-83242009000500007. PMID 19838557
- [Background] Tsai TH, Tsai TH, Chien YC, Lee CW, Tsai PJ. In vitro antimicrobial activities against cariogenic streptococci and their antioxidant capacities: A comparative study of green tea versus different herbs. Food Chem. 2008 Oct 15;110(4):859-64. doi: 10.1016/j.foodchem.2008.02.085. Epub 2008 Mar 4. PMID 26047271
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Derived] Abdulbaqi HR, Himratul-Aznita WH, Baharuddin NA. Evaluation of Salvadora persica L. and green tea anti-plaque effect: a randomized controlled crossover clinical trial. BMC Complement Altern Med. 2016 Dec 1;16(1):493. doi: 10.1186/s12906-016-1487-0. PMID 27903262